CLINICAL TRIAL: NCT02092545
Title: Heart Obesity Prevention Education: Retired NFL Players Weight Management Study
Brief Title: Heart Obesity Prevention Education
Acronym: HOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampa General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGH0002
Record Dates: First submitted 2014-03-13; First posted 2014-03-20 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketogenic diet (Other): Weight management on a male population of retired NFL athletes.
  Interventions: Other: Ketogenic diet

INTERVENTIONS:
Other: Ketogenic diet
  Other Names: High protein; Low carbohydrate

SUMMARY:
Study to collect data on weight management on a male population of retired NFL athletes.

DETAILED DESCRIPTION:
Up to ten retired NFL players will receive a comprehensive and monitored weight loss program using a protocol that has been established at the TGH+USF Bariatric Center. A low calorie diet with meal replacements will be used and over the course of the study the participants will be taught to eat low calorie nutritious foods. The sessions will teach proper eating habits, stress control, and skills to maintain a healthy weight.

The length of the study is 6 months. Treatment will last 24 weeks, the participants will attend group sessions (60-90 mins.) on a weekly basis for weeks 1-12 and then every other week for weeks 14-24, for a total of 18 treatments. Treatment will include meal replacement, education on nutrition and proper eating habits as well as behavior modification and skills which is known to be effective.

Participants will be scheduled to come to the Bariatric Center for the first assessment/screening and for the consenting process. TGH+USF Bariatric Center has dedicated clinical space in their suite with private exam rooms, an education classroom, and private testing room.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Former NFL players
* Aged 25-64 (Age range is chosen to keep participants as uniform as possible given the small number of participants. The majority of the players are in this age range and participants need to be able to exercise and be active. Also the NFL in its current form was created in 1970 so there are very few players that are retired from the NFL that are over the age of 65.)
* BMI >27
* English- speaking

Exclusion Criteria:

* Cancer within the last 5 years (except non-melanoma skin cancer)
* Significant Cardiovascular Disease (recent < 1 year Myocardial Infarction, hospital admission < 1year for Congestive Heart Failure, Active Angina, exercise induced Angina)
* Malignant arrhythmias (VTACH, AFIB, Aflutter)
* Renal Disease ( Dialysis or Chronic Renal Insufficiency)
* Hepatic Disease ( Hepatitis B and C or Liver function test 2.5 times the upper limits of normal, or liver transplant that requires immune odulating/suppressing medications, ammonia lowering medications, or hepatic disease related to diet modification).
* Psychosis, Severe Anxiety, or Major Depression
* Significant migraines requiring abortive medication in the last year
* Significant Endocrine dysfunction ( Cushing's Syndrome )
* Uncontrolled Hypertension > 160/90
* Severe arthritis that significantly limits mobility
* Uncontrolled Hyper/Hypothyroidism
* Obesity Surgery in the past
* Weight loss of greater than 10% of the subjects body weight in the last year
* Recent history (within 1 year ) of Alcohol abuse, illegal Drug abuse
* Active pulmonary disease that requires daily corticosteroids, an oxygen requirement, or ventilation support for chronic disease management.
* Participants currently taking or having been taking within the last 3 months the following medication will be excluded.
* Appetite Suppressants (Phenterimine, Qsymia)
* Anti-obesity medications (Xenical/Meridia)
* Corticosteroids or > 1500 micrograms of inhaled steroids daily
* Raloxifene (Evista) or Temoxifene (HRT medications)
* Inappropriate use of Testosterone
* At the discretion of the investigator use of Psychiatric Medication, Sedative/Hypnotics, Benzodiazepines
* Detailed Disease and Lab Value Exclusion
* Active rheumatologic, dermatologic disease, or autoimmune/inflammatory condition will be defined as any patient who currently, or has a past medical history of chronic (>2 weeks) immune modulating/suppressing medications.
* Active renal disease will be defined as any patient who is currently, or has a history requiring potassium phosphate lowering medication, protein restriction diet, or hemo/peritoneal dialysis
* Screening creatinine >1.5
* Serious or unstable medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
* Participants with screening triglycerides above 500 mg.
* Uncontrolled Dyslipidemia as defined by screening LDL cholesterol >160 mg/dL. Participants on medication treating dyslipidemia for at least 3 months are allowable.
* Neuropathy that interferes with exercise.
* Previous weight loss surgery
* Lab value exclusions are limited to all routine electrolyte values outside the normal range, except glucose.

Ages: 25 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in body mass index from start of study in 6 month timeframe. | 6 months
  Calculate change in weight and BMI

CONTACTS AND LOCATIONS:
Overall Officials: John Gonzalvo, DO, Principal Investigator — Tampa General Hospital
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States